CLINICAL TRIAL: NCT02690220
Title: National, Multicentre Post Market Surveillance Study on Anterior Pelvic Prolapse Reconstruction With a Titanium-coated Polypropylene Mesh (TiLOOP® PRO A)
Brief Title: Anterior Pelvic Prolapse Reconstruction With TiLOOP® PRO A Polypropylene Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: pfm medical gmbh (Industry)
Collaborators: Crolll Gmbh (Other); Bayes GmbH (Other); Aix Scientifics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pfm15k001 TiLOOP® PRO A
Record Dates: First submitted 2016-02-05; First posted 2016-02-24 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-01

CONDITIONS: Cystocele; Uterine Prolapse
Keywords: polypropylene mesh; prolapse; cystocele; surgical mesh
MeSH Terms: conditions — Cystocele; Uterine Prolapse; Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgical mesh implantation (Other): Standard method to implant the TiLOOP® PRO A surgical mesh transvaginally. Women with a symptomatic genital descensus: at least stage II (ICS-classification according Pelvic Organ Prolapse Quantification System (POP-Q system)). This applies to primary as well as recurrent intervention.
  Interventions: Device: TiLOOP® PRO Plus A

INTERVENTIONS:
Device: TiLOOP® PRO Plus A — The standard operation method for the surgical repair of anterior prolapse is via the obturator membrane. The mesh is placed trans-vaginally using the TiLOOP® Application Set to place the mesh arms.

SUMMARY:
The purpose of this study is to determine the influence of anterior pelvic prolapse reconstruction with a titanized polypropylene mesh on patients quality of life.

DETAILED DESCRIPTION:
This multicentre, non-randomized, observational clinical investigation will be performed to obtain usability and postmarket information on the TiLOOP® pelvic floor reconstruction meshes and in particular to obtain the improvement of patients' quality of life.

It is expected that the patient's quality of life is meliorated after implantation of a TiLOOP® PRO A mesh. To verify this, it will be shown that by means of a validated questionnaire the subjective quality of life after 12 months is significantly better than before implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Existence of a cystocele. Women with a symptomatic genital descensus: at least stage II (ICS-classification according POP-Q system). This applies to primary as well as recurrent intervention.
2. Patient is mentally able to understand the nature, aims, or possible consequences of the clinical investigation.
3. Patient information has been handed out and written consent is at hand.
4. Patient has attained full age (18 years or older).

Exclusion Criteria:

1. Unfinished family planning, pregnancy or breast-feeding mother.
2. Known intolerance to the mesh-implants under investigation.
3. Lack of written patients' informed consent.
4. Lack of patient compliance regarding data collection, treatment or follow-up investigations in the scope of the protocol.
5. Patients with acute (within the last 12 months) carcinoma in the pelvic area.
6. Patients with history of radiotherapy in the pelvic area.
7. Patients with implanted anterior pelvic floor mesh.
8. Patient is institutionalized by court or official order (MPG §20.3).
9. Participation in another interventional clinical investigation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Patient's Quality of Life | 12 months
  By means of a validated questionnaire it will be shown whether the subjective quality of life after 12 months is significantly better than before implantation.

SECONDARY OUTCOMES:
Patient's Quality of Life | 6 months
  The evaluation of changes in quality of life assessed by the P-QoL 6 months after implantation of the TiLOOP® PRO A surgical mesh compared to before implantation.
Adverse Events (AE) | 6 weeks, 6 and 12 months
  Assessment and analysis of all [serious] adverse events ([S]AEs) during the first 12 months after implantation along with a contextual placement of safety data based on current literature.
Feasibility Check of Mesh implantation | 1 day
  To evaluate mesh implantation, information about the duration of the procedure (minutes from cut to stitches) and the operability of the application set (easy, suitable, difficult, no set used) will be collected during the surgery. Taking together, this information will encapsulate the feasibility of the mesh implantation descriptively.
Number of complications and concomitant procedures | 1 day
  Counting the number of intraoperative complications (e. g. lesion of the bladder, the urethra or the intestines) and concomitant procedures (e. g. hysterectomy, colporrhaphy, vaginal sacrospinal fixation) procedure-related adverse events as assessed by CTCAE v4.0 and common concomitant procedures will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fünfgeld, Dr. med., Principal Investigator — Klinik Tettnang GmbH
Locations (5):
- Germany (5):
  - Klinik Tettnang GmbH, Tettnang, Baden-Wurttemberg
  - Klinikum Augsburg, Augsburg, Bavaria
  - Klinikum Dresden-Friedrichstadt, Dresden, Saxony
  - Klinikum Oberlausitzer Bergland gemeinnützige GmbH, Zittau, Saxony
  - Ev. Amalie-Sieveking-Krankenhaus, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cadenbach-Blome T, Grebe M, Mengel M, Pauli F, Greser A, Funfgeld C. Significant Improvement in Quality of Life, Positive Effect on Sexuality, Lasting Reconstructive Result and Low Rate of Complications Following Cystocele Correction Using a Lightweight, Large-Pore, Titanised Polypropylene Mesh: Final Results of a National, Multicentre Observational Study. Geburtshilfe Frauenheilkd. 2019 Sep;79(9):959-968. doi: 10.1055/a-0984-6614. Epub 2019 Sep 11. PMID 31523096